CLINICAL TRIAL: NCT06728917
Title: Occult Hepatitis B Virus Infection and HBV Reactivation After Switching to Long Acting Therapy in Patients Living With HIV-1
Brief Title: Occult Hepatitis B Virus Infection and HBV Reactivation After Switching to Long Acting Therapy in Patients With HIV-1
Acronym: OBILART
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Università Luigi Vanvitelli della Campania (Unknown)
Responsible Party: Principal Investigator, Castagna Antonella, Prof, IRCCS San Raffaele
Other Study IDs: IRCCS San Raffaele
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: HBV (Hepatitis B Virus); HIV Infection
Keywords: Occult hepatitis B virus infection; long acting therapy; people living with HIV-1; HBV reactivation
MeSH Terms: conditions — Hepatitis B; HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collection at baseline (start of long-acting therapy) weeks 12, 24 and 48 after the start of long-acting therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects living with HIV switching to long acting therapy: The study will include subjects living with HIV, followed at the San Luigi Center (Infectious Diseases), IRCCS Ospedale San Raffaele in Milan, Integrated Infectious Risk Management Department, Policlinico S. Orsola-Malpighi in Bologna, and the Department of Mental and Physical Health and Medicine prevention, University of Campania L. Vanvitelli of Naples, who agree to the switch from the current antiretroviral regimen which includes drugs active on HIV/HBV to long acting therapy.

SUMMARY:
The primary objective of the present project will be to investigate the risk of HBV reactivation (from virological reactivation to overt HBV infection) in HIV-1 carriers with occult HBV infection (OBI, is characterized by the absence of surface antigenemia, HBsAg negativity, with the presence of HBV-core antibody, HBcAb) and switching from antiretroviral therapy (ART) including nucleos(t)ides to long-acting formulation.

DETAILED DESCRIPTION:
Observational prospective, multicenter, single-arm study with additional procedure in people living with HIV-1 and having serological markers of previous HBV infection: anti-core antibodies and/or antibodies against surface antigen (HBsAb) and switching from nucleoside analogue therapy to long-acting therapy including cabotegravir (CAB, HIV-1 integrase inhibitor) + rilpivirine (RPV, non-nucleoside HIV-1 reverse transcriptase inhibitor) intramuscularly 1 time every 2 months.

Primary Objective To study the risk of HBV reactivation from the phase of possible virological reactivation (HBV-DNA >=10 IU/mL), when the liver enzymes are within normal limits to overt HBV infection. Overt HBV infection is characterized by positive HBV-DNA, possible positivity of surface antigen (HBsAg) with or without altered liver enzymes in HIV-1 patients with OBI, with switch from ART, which includes nucleos(t)ide analogues active on the two HIV/HBV viruses, to the long-term formulation in which nucleos(t)ide analogues active on the two viruses are not included.

Secondary Objectives

* To evaluate the effect, in the context of HBV reactivation, of HBV-RNA as a surrogate marker of the transcriptional activity of the covalently closed circular (cccDNA) which is present as an HBV replication intermediate at the hepatocyte level.
* Examine the mutational profile of HBV domains (pre-S1 and S genes, X gene), mutations in the nucleocapsid promoter region and the pre-core/core variant, capable of influencing HBV replication efficiency, including also the analysis of mutants characterized as viral escape.

Exploratory Objectives To study the mutational profile of the regions of the hepatitis B virus (HBV) able to influence replication efficiency.

The study will include subjects living with HIV, followed at the San Luigi Center (Infectious Diseases), IRCCS Ospedale San Raffaele in Milan, Integrated Infectious Risk Management Department, Policlinico S. Orsola-Malpighi in Bologna, and the Department of Mental and Physical Health and Medicine prevention, University of Campania L. Vanvitelli of Naples, who agree to the switch from the current antiretroviral regimen which includes drugs active on HIV/HBV to long acting therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Informed consent to participate in the study
* HIV infection
* Stable antiretroviral therapy (ART) in the six months prior to enrollment without virological failure defined by HIV-RNA>50 copies/mL in at least two consecutive determinations
* Positive HBV anti-core antibodies (HBcAb) in the absence of hepatitis B surface antigen (HBsAg)
* Absence of mutations associated with resistance to integrase inhibitors (INSTIs) and reverse transcriptase inhibitors (NNRTIs) by HIV genotypic resistance testing
* CD4 Nadir >200 cells/mm3

Exclusion Criteria:

* Any contraindications to the use of one or more long-acting drugs
* Non-expression or withdrawal of informed consent to participate in the study
* Pregnancy
* Lack of HIV genotypic resistance testing
* Virological failure (HIV-RNA >50 copies/mL in at least 2 consecutive determinations) in the 6 months prior to enrollment
* Therapeutic interruptions in the six months prior to enrollment, excluding interruptions lasting less than a month due to tolerability
* CD4 Nadir =<200 cells/mm3
* Presence of biochemical signs of hepatocellular necrosis (AST, ALT > normal values as indicated in laboratory tests).
* Cirrhosis and/or fibrosis score >F3 assessed by transient elastography (FibroScan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 subjects will participate to the study, 30 subjects enrolled at the San Luigi Center (Unit of Infectious Diseases), IRCCS Ospedale San Raffaele in Milan, 10 subjects enrolled at Integrated Infectious Risk Management Department, Policlinico S. Orsola-Malpighi in Bologna, and 10 at the Department of Mental and Physical Health and Medicine prevention, University of Campania L. Vanvitelli of Naples.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Quantification of hepatitis B DNA (HBV-DNA) | Baseline (start of long-acting therapy) weeks 12, 24 and 48
  HBV-DNA increase respect to baseline viremia (=>10 IU/mL) according to different time points (W12, W24, W48) after the start of LART.

SECONDARY OUTCOMES:
Quantification of hepatitis B RNA (HBV-RNA) | Baseline and at weeks 12, 24 and 48
  any concomitant HBV-RNA increase respect to baseline value by measurement of HBV- RNA at different time points (W12, W24, W48).
HBV mutational pattern by direct sequencing (Sanger) | Baseline and at weeks 12, 24 and 48
  the mutational pattern of HBV genome (S, pre-C/C, X and polymerase regions) will be evaluated in positive HBV-DNA samples

OTHER OUTCOMES:
Measurement of number of amino acid and/or nucleotide substitution. | Baseline (start of long-acting therapy) weeks 12, 24 and 48
  Measurement of number of amino acid and/or nucleotide substitution tostudy the mutational profile of the regions of the hepatitis B virus (HBV) able to influence replication efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Castagna, Prof, MD, Principal Investigator — IRCCS San Raffaele
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - IRCCS San Raffaele O.U. Infectious Diseases, Milan
  - Università Luigi Vanvitelli della Campania, Napoli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morsica G, Bagaglio S, Cicconi P, Capobianchi MR, Pellizzer G, Caramello P, Orani A, Moioli C, Rizzardini G, Uberti-Foppa C, Puoti M, Monforte AD; Hepa I.C.o.N.A the Icona Foundation Study Groups. Viral interference between hepatitis B, C, and D viruses in dual and triple infections in HIV-positive patients. J Acquir Immune Defic Syndr. 2009 Aug 15;51(5):574-81. doi: 10.1097/QAI.0b013e3181add592. PMID 19590432
- [Background] Jaeger H, Overton ET, Richmond G, Rizzardini G, Andrade-Villanueva JF, Mngqibisa R, Hermida AO, Thalme A, Belonosova E, Ajana F, Benn PD, Wang Y, Hudson KJ, Espanol CM, Ford SL, Crauwels H, Margolis DA, Talarico CL, Smith KY, van Eygen V, Van Solingen-Ristea R, Vanveggel S, Spreen WR. Long-acting cabotegravir and rilpivirine dosed every 2 months in adults with HIV-1 infection (ATLAS-2M), 96-week results: a randomised, multicentre, open-label, phase 3b, non-inferiority study. Lancet HIV. 2021 Nov;8(11):e679-e689. doi: 10.1016/S2352-3018(21)00185-5. Epub 2021 Oct 11. PMID 34648734
- [Background] Huang H, Wang J, Li W, Chen R, Chen X, Zhang F, Xu D, Lu F. Serum HBV DNA plus RNA shows superiority in reflecting the activity of intrahepatic cccDNA in treatment-naive HBV-infected individuals. J Clin Virol. 2018 Feb-Mar;99-100:71-78. doi: 10.1016/j.jcv.2017.12.016. Epub 2018 Jan 6. PMID 29353073
- [Background] Carey I, Gersch J, Wang B, Moigboi C, Kuhns M, Cloherty G, Dusheiko G, Agarwal K. Pregenomic HBV RNA and Hepatitis B Core-Related Antigen Predict Outcomes in Hepatitis B e Antigen-Negative Chronic Hepatitis B Patients Suppressed on Nucleos(T)ide Analogue Therapy. Hepatology. 2020 Jul;72(1):42-57. doi: 10.1002/hep.31026. PMID 31701544
- [Background] Bagaglio S, Bianchi G, Danise A, Porrino L, Uberti-Foppa C, Lazzarin A, Castagna A, Morsica G. Longitudinal evaluation of occult hepatitis B infection in HIV-1 infected individuals during highly active antiretroviral treatment interruption and after HAART resumption. Infection. 2011 Apr;39(2):121-6. doi: 10.1007/s15010-011-0093-9. Epub 2011 Mar 22. PMID 21424854
- [Background] Bagaglio S, Porrino L, Lazzarin A, Morsica G. Molecular characterization of occult and overt hepatitis B (HBV) infection in an HIV-infected person with reactivation of HBV after antiretroviral treatment interruption. Infection. 2010 Oct;38(5):417-21. doi: 10.1007/s15010-010-0032-1. Epub 2010 Jun 9. PMID 20533073
- [Background] Clark SJ, Creighton S, Horner M, Smith HM, Portmann B, Taylor C, Cramp ME. Reactivation of latent hepatitis B virus infection with HIV-related immunosuppression. Int J STD AIDS. 2006 Jan;17(1):67-9. doi: 10.1258/095646206775220612. PMID 16409685
- [Background] Chamorro AJ, Casado JL, Bellido D, Moreno S. Reactivation of hepatitis B in an HIV-infected patient with antibodies against hepatitis B core antigen as the only serological marker. Eur J Clin Microbiol Infect Dis. 2005 Jul;24(7):492-4. doi: 10.1007/s10096-005-1355-1. PMID 15990987
- [Background] Onorato L, Pisaturo M, Camaioni C, Grimaldi P, Codella AV, Calo F, Coppola N. Risk and Prevention of Hepatitis B Virus Reactivation during Immunosuppression for Non-Oncological Diseases. J Clin Med. 2021 Nov 8;10(21):5201. doi: 10.3390/jcm10215201. PMID 34768721
- [Background] Hu KQ. Occult hepatitis B virus infection and its clinical implications. J Viral Hepat. 2002 Jul;9(4):243-57. doi: 10.1046/j.1365-2893.2002.00344.x. PMID 12081601
- [Background] Mulrooney-Cousins PM, Michalak TI. Persistent occult hepatitis B virus infection: experimental findings and clinical implications. World J Gastroenterol. 2007 Nov 21;13(43):5682-6. doi: 10.3748/wjg.v13.i43.5682. PMID 17963292
- [Background] Ramezani A, Mohraz M, Aghakhani A, Banifazl M, Eslamifar A, Khadem-Sadegh A, Velayati AA. Frequency of isolated hepatitis B core antibody in HIV-hepatitis C virus co-infected individuals. Int J STD AIDS. 2009 May;20(5):336-8. doi: 10.1258/ijsa.2008.008377. PMID 19386971
- [Background] Pisaturo M, Onorato L, Russo A, Coppola N. Prevalence of occult HBV infection in Western countries. J Med Virol. 2020 Dec;92(12):2917-2929. doi: 10.1002/jmv.25867. Epub 2020 Jun 29. PMID 32275083
- [Background] Santos EA, Yoshida CF, Rolla VC, Mendes JM, Vieira IF, Arabe J, Gomes SA. Frequent occult hepatitis B virus infection in patients infected with human immunodeficiency virus type 1. Eur J Clin Microbiol Infect Dis. 2003 Feb;22(2):92-8. doi: 10.1007/s10096-002-0868-0. Epub 2003 Feb 18. PMID 12627282
- [Background] Nunez M, Rios P, Perez-Olmeda M, Soriano V. Lack of 'occult' hepatitis B virus infection in HIV-infected patients. AIDS. 2002 Oct 18;16(15):2099-101. doi: 10.1097/00002030-200210180-00024. No abstract available. PMID 12370518
- [Background] Raimondo G, Pollicino T, Cacciola I, Squadrito G. Occult hepatitis B virus infection. J Hepatol. 2007 Jan;46(1):160-70. doi: 10.1016/j.jhep.2006.10.007. Epub 2006 Nov 7. PMID 17112622